CLINICAL TRIAL: NCT01163383
Title: I-Metaiodobenzylguanidine (131 I-MIBG) Therapy for Refractory Neuroblastoma, Expanded Access Protocol
Brief Title: 131-I-MIBG Therapy for Refractory Neuroblastoma, Expanded Access Protocol
Status: Available | Type: Expanded Access
Sponsor: John Maris (Other)
Responsible Party: Sponsor-Investigator, John Maris, Director of Children's Hospital Cancer Center, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Other Study IDs: 05-004159; CHP-830 (Other: The Children's Hospital of Philadelphia)
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma; Childhood Metastatic Pheochromocytoma
Keywords: Refractory Neuroblastoma; Recurrent Neuroblastoma; Neuroblastoma; stage IV neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine

INTERVENTIONS:
Drug: 131 I-Metaiodobenzylguanidine (131 I-MIBG) — 131 I-MIBG 1-18mCi/kg given intravenously on day 1. Subjects may receive multiple courses every 4-8 weeks depending on the dose given.
  Other Names: MIBG; 131 I-Metaiodobenzylguanidine; radioactive Iodine (131); Metaiodobenzylguanidine
Drug: 131 I-MIBG — 131-I-MIBG will be infused intravenously over 60-90 minutes once per course. The dose will be determined by the treating physician.
  Other Names: 131 I- Metaidobenzylguanidine; MIBG; Radioactive iodine; Metaiodobenzylguanidine therapy

SUMMARY:
Metaiodobenzylguanidine (MIBG) is a substance that is taken up by neuroblastoma cells. MIBG is combined with radioactive iodine (131 I) in the laboratory to form a radioactive compound 131 I-MIBG. This radioactive compound delivers radiation specifically to the cancer cells and causes them to die.

The purpose of this research protocol provides a mechanism to deliver MIBG therapy when clinically indicated, but also to provide a mechanism to continue to collect efficacy and toxicity data that will be provided.

A recent New Approaches to Neuroblastoma Therapy (NANT) phase 2 randomized trial of 131I-MIBG with or without radiation sensitizers for relapsed refractory or persistent neuroblastoma enrolled 114 patients ages 1-30 years showed that Arm A (MIBG alone) had a response rate of 17%, Arm B (MIBG with Vincristine and Irnotecan) had a response rate of 14% and Arm C (MIBG with vorinostat) had a response rate of 32% after the first cycle. After the second cycle, Arm A had a response rate of 33%, Arm B had 30% response rate and Arm C had a 75% response rate. There was an excess of toxicities in Arm B, and no significant SAEs in Arm C. These data were reported at the American Society of Clinical Oncology meeting in June of 2020.

Vorinostat has been used extensively in adults and has been granted US FDA approval for the treatment of cutaneous T-cell lymphoma. The approved adult dose is 400 mg orally once daily. Vorinostat is not FDA approved for use in neuroblastoma.

DETAILED DESCRIPTION:
131I-MIBG is experimental, but has been used in more than 100 children in the United States by itself to treat relapsed neuroblastoma. A recent study using increasing doses of 131I-MIBG in both children and adults with relapsed neuroblastoma or metastatic pheochromocytoma/ganglioma showed anti-cancer effects in some of these patients. The main side effect of this treatment was a decrease in the number of normal blood-forming cells (called stem cells) in the bone marrow, but a dose of 12 mCi/kg did not cause permanent damage to the bone marrow in a small number of patients.

There are certain tests or procedures that will need to be done to confirm that the subject is eligible for this therapy. These include lab work, physical exam and MIBG scan. A CT scan, an MRI, a bone scan, bone marrow aspirate and biopsy and urine tests will be done to evaluate your disease status when clinically indicated. Your doctor will determine which tests are required.

Subjects will need to have an intravenous catheter (tube) placed in a vein before beginning study treatment. An existing central venous catheter can be used to administer the medicine.

Because subjects' urine will be radioactive, a urinary catheter may be inserted to ensure drainage of the urine, which will be radioactive. The catheter will be removed 3-5 days following the treatment. General anesthesia or sedation is typically given for the procedure of inserting the catheter.

Subjects will be treated in a specially prepared room in the CHOP Pediatric Oncology Unit. Upon admission, the nursing staff will instruct caregivers on the care of the subject following the MIBG infusion. Because of the frequent exposure of the nursing staff to radiation and the high level of radiation surrounding the subject during therapy, the nurses' contact will be limited to complex medical care, so that they are available for subjects in the event of an emergency. Adult family members will be expected to be present at all times during the hospitalization to:

* Assist with hygiene
* Give oral medications
* Offer and empty bedpans
* Assist with meals
* Change diapers (if used)
* Change clothing and bed linens if soiled
* Entertain or distract individuals who become upset or restless due to the isolation or procedures.
* Record Dosimeter readings.

Isolation: For 2-5 days subjects will be placed in a single room with a bed surrounded by lead shielding to prevent exposure of visitors and hospital personnel to radioactivity. Family members may visit in the room, but must wear a radiation badge to measure exposure. A single family member can sleep in the room, but no one is allowed to go behind the shields or sleep in the bed with the child.

Subjects will receive fluids through the central venous catheter. The fluids will begin at least four hours before and continue at least 72 hours after the 131I-MIBG treatment begins.

Subjects will take a medicine by mouth, potassium iodide, to prevent thyroid damage from the radioactive iodine contained in the 131I-MIBG. This medication will be taken on the day of the treatment and will continue for a total of 6 weeks.

The 131I-MIBG will be given through an intravenous catheter over 1-2 hours.

During the administration of the drug, subject's blood pressure and heart rate will be checked frequently.

Before and at regular intervals after treatment, subjects will have routine blood tests to check his/her blood counts, hormone, liver and kidney functions. Blood will be checked frequently for the first 1-6 weeks, and 6 weeks after the treatment. Approximately 1 teaspoon of blood will be drawn each time during the first 6 weeks to perform the tests listed above.

An MIBG scan will be performed to see where the drug is concentrating in the body following treatment. No injection of a radioactive marker will be required and this is usually done on the day for discharge. It is identical to the pretherapy MIBG scan except for not needing MIBG injection and it is usually shorter (15-30 minutes).

Six to eight weeks after treatment, an MIBG and other scans will be done to evaluate the response of the tumor to the treatment.

If the subject's tumor is responding or stable 6-7 weeks after each treatment, they may be eligible for a second and third course of treatment, as long as their white blood counts have recovered from the treatment and the patient has stem cells available if needed. If another MIBG treatment is given, it will be at the same dose as the first treatment, unless it is thought to be necessary for safety reasons (based on toxicity information from the first infusion) to decrease the dose.

If the subject's blood counts decrease following the therapy, treatment with Filgrastim (G-CSF) or Neulasta may be required. G-CSF/neulasta is a medicine that helps increase the white blood cells. This is given by a subcutaneous (under the skin) injection (like an insulin shot). GCSF is given daily and Neulasta is given every 14 days instead of GCSF. Neulasta works like GCSF to help increase the white blood counts but lasts longer in your child's body. This medicine will start if the absolute neutrophil count (ANC), a measure of the infection fighting cells, goes below 500 and will continue until recovery, generally above 5000.

Vorinostat may be given at the discretion of the PI and treating physician as a clinical procedure. This will be administered for clinical purposes, regardless of study participation. Patients will receive 180 mg/m2/dose (maximum dose 400 mg) as in the recently completed NANT study once daily by mouth, NG, or G-tube on days -1 to +12 (14 total doses). Vorinostat will be given for 14 days continuously. Vorinostat should be taken with food or within 30 minutes after a meal. The dose should be taken in the morning whenever possible. On day 1 of therapy, vorinostat should be taken 1 hour prior to the start of the 131I-MIBG infusion.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed neuroblastoma
* Age greater than 1 year.
* Performance Level: Patients must have a Karnofsky or Lansky performance status of equal to or greater than 50 percent
* Disease status: Failure to respond to standard therapy (usually combination chemotherapy with or without radiation and surgery) or development of progressive disease at any time. Disease evaluable by MIBG scan must be present within 8 weeks of study entry and subsequent to any intervening therapy. The principal or co-investigator can waive the requirement for intervening therapy if in their judgment this would pose undue risk and would not affect ability to judge treatment effectiveness.
* Stem cells: Patients must have a hematopoietic stem cell product available for re-infusion after MIBG treatment at doses of >/= 12 mCi/kg. The recommended minimum quantity for peripheral blood stem cells based on documentation from the time of collection is 1.0 x 10^6 CD34+ cells/kg. The minimum dose for bone marrow is 1.0 x 10^8 mononuclear cells/kg. If no stem cells are available, the dose of 131I-MIBG should be ≤ 12 mCi/kg.
* Prior Therapy: Patients may enter this study with or without re-induction therapy for recurrent tumor. Patients must have fully recovered from the toxic effects of any prior therapy. Subjects cannot be receiving chemotherapy, cytokine therapy or other investigational agents, and must have fully recovered from the toxic effects of any prior therapy. No investigational agents are allowed in this time frame, but FDA-approved drugs for other indications that are not cytotoxic are allowed to be used off label if this is considered in the best interest of the patient by the investigator. No concomitant cytotoxic therapy is permitted with the exception of vorinostat.
* Liver function: Bilirubin ≤2x upper limit of normal; AST/ALT ≤10x upper limit of normal
* Kidney function: Creatinine ≤3x upper limit of normal
* Signed informed consent: The patient and/or the patient's legally authorized guardian must provide written informed consent to participate in this expanded access protocol.

Exclusion criteria

* Patients with disease of any major organ system that would compromise their ability to withstand therapy, as deemed by the principal investigator or treating sub-investigator.
* Because of the teratogenic potential of the study medications, no patients who are pregnant or lactating will be allowed. Patients of childbearing potential must practice an effective method of birth control while participating on this study, to avoid possible damage to the fetus.
* Patients who are on hemodialysis
* Patients with uncontrolled infections
* Exceptions to the above eligibility criteria may be allowed if approved by the principal investigator as long as exception does not compromise the safety of the subject and the exception is clearly documented. Each protocol exception must be reviewed by the Institutional Review Board before therapy is initiated.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John M Maris, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States